CLINICAL TRIAL: NCT03002597
Title: Visual Information Restoration and Rehabilitation Via Sensory Substitution Technology in Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Issue reaching target enrollement
Sponsor: Ellen Mitchell (Other)
Responsible Party: Sponsor-Investigator, Ellen Mitchell, Assistant Professor of Ophthalmology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19080134
Record Dates: First submitted 2016-12-20; First posted 2016-12-26 (Estimated); Results first posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-07

CONDITIONS: Blindness
MeSH Terms: conditions — Blindness

ARMS (2):
- Blind Children (Experimental): Children between the ages of 4 and 17 who are blind (documented visual acuity of light perception or worse) in both eyes from an eye care provider.
  Interventions: Device: BrainPort V200 Device
- Sighted Children (Experimental): Children between the ages of 4 and 17 who are sighted in both eyes.
  Interventions: Device: BrainPort V200 Device

INTERVENTIONS:
Device: BrainPort V200 Device — To see if the device can be used in a pediatric population by measuring the subjects' improvement over baseline in any of the following areas: light detection, light localization, movement perception, and standardized object recognition tasks after use of the BrainPort.

SUMMARY:
The BrainPort vision device is a visual prosthetic designed for those who are blind. It enables perception of visual information using the tongue and camera system as a paired substitute for the eye. Visual information is collected from a video camera and translated into a gentle vibration that is presented to the subject on the tongue. With training users perceive shape, size, location and motion of objects in their environment. It is a functional, non-surgical device developed to demonstrate as an aid to the visually impaired.

The aim of this proposal is to evaluate a non-surgical visual prosthetic (BrainPort vision device) that enables the blind to appreciate their immediate surroundings and determine the way the brain interprets the information. Our goal is to determine if the device can be used in a pediatric population by measuring the subjects' improvement over baseline in any of the following areas: light detection, light localization, movement perception, and standardized object recognition tasks after use of the BrainPort.

DETAILED DESCRIPTION:
Objective:

Our objective is to determine if the functional improvements seen in blind subjects using the BrainPort can be realized in a pediatric cohort.

Specific Aims:

The aim of this proposal is to evaluate a non-surgical visual prosthetic (BrainPort vision device) that enables the blind to appreciate their immediate surroundings and determine the way the brain interprets the information. Our main goal is to determine if the device can be used in a pediatric population by measuring the subjects' improvement over baseline in any of the following areas: light detection, light localization, movement perception, and standardized object recognition tasks after use of the BrainPort.

As a second aim, the investigators will use a multimodal MR scanning session to study the neurophysiological basis of sensory substitution in children. Under this aim the investigators will pursue two main objectives. First, the investigators will correlate the behavioral data with the imaging data in order to detect regions of the brain where structure and/or function are associated with successful use of sensory substitution devices. Second, the investigators will utilize these data along with previously collected adult data to model the effects of prior visual experience on visual cortex plasticity due to blindness.

Background:

The BrainPort vision device is a visual prosthetic designed for those who are blind. It enables perception of visual information using the tongue and camera system as a paired substitute for the eye. Visual information is collected from a video camera and translated into gentle electrical stimulation patterns on the surface of the tongue. With training, users perceive shape, size, location and motion of objects in their environment. It is a functional, non-surgical device developed to demonstrate as an aid to the visually impaired.

Tactile sensory systems have proven capable of carrying information to the brain that is usually acquired visually. Braille and the long cane have provided such information to blind persons for decades, and in the 1960's it was clearly demonstrated that tactile inputs could provide access to written print1 and visual images2. The main limitation to the development of practical vision substitution has been the inadequacy of brain-machine interfaces. Thirty-five years ago Paul Bach-y-Rita, MD wrote "That a successful sensory substitution system is not presently in use may not be due to limited functional capabilities of the brain; it may be due to the fact that an artificial receptor system has not yet been constructed to challenge the adaptive capacities of the human brain"3.

BrainPort Vision Device Since 1998, Wicab has focused on biomedical engineering research and development of commercial devices based on its proprietary BrainPort® technology4. The BrainPort vision device is a visual prosthetic designed for those who are blind.

Numerous previous studies support using the tongue as a sensory substitution channel2,3,5-8. Our and others' research has revealed that the brain can correctly interpret information from a sensory substitution device, even when the information is not presented in the same pathway as the natural sensory system. For example, the optical image actually received by the eye travels no farther than the retina, which converts the image into spatio-temporal patterns of action potentials along the optic nerve fibers. By analyzing these impulse patterns, the brain recreates the image. These impulses are not unique for vision. In fact, all sensory systems code information using the same 'language': neuronal action potentials. Using the vision example as a paradigm, sensory substitution requires only that action potentials be accurately entrained in the alternate sensory information channel. With training, the brain may learn to appropriately interpret information from the alternate channel and then to process that information much as it would data from the intact natural sense. Therefore, this technology benefits users by stimulating the tongue with usable information about their environment, which some users have described as resembling vision.

Although BrainPort technology stimulates the tongue through the electrode array, the stimulation is not at all painful; a BrainPort device emits only 11.85 µJ per pulse (regulatory limit for cutaneously electrical stimulating devices: 300 mJ). In fact, users often report the sensation as being like champagne bubbles effervescing on the tongue. Participants using BrainPort devices, whether for several hours each day over the course of a few weeks or for 20 minutes a day for up to one year, report no discomfort.

Little work has been done using imaging to study blind children. Werth and Seelos used fMRI to measure evoked activity in the visual cortex of children as evidence of visual function improvement following field training (Neurpsychologica. 2005. 43(14): 2011). However, to our knowledge, imaging of blind children to assess plasticity of the visual cortex at such a young age has not been done. In the short term, imaging of these subjects may improve our ability to screen for patients who would benefit from sensory substitution devices as well as to evaluate training paradigms. In the long term, understanding plasticity due to visual deprivation will be important not just for sensory substitution, but for all vision restoration strategies in order to identify subjects still capable of processing visual input. As the investigators attempt to model the effects of prior visual experience on plasticity in the visual cortex following blindness, children represent a unique and essential portion of the sample to tease apart the relative effects of blindness duration and early versus late acquisition.

The BrainPort device has been approved by the FDA since June of 2015.

Significance:

The BrainPort vision device is a visual prosthetic designed for those who are blind. It enables perception of visual information using the tongue and camera system as a paired substitute for the eye. Visual information is collected from a video camera and translated into gentle electrical stimulation patterns on the surface of the tongue. With training users perceive shape, size, location and motion of objects in their environment. It is a functional, non-surgical device developed to demonstrate as an aid to the visually impaired. The BrainPort vision device is the only new technology likely available in the near term to address safety and mobility issues resulting from blindness.

Our results have shown that the use of the BrainPort results in behavioral improvements as well as activation in visual cortical regions using fMRI and PET scans in adults. A trial which seeks to determine if functional abilities can also be improved in a pediatric cohort is justifiable for the following reasons:

1. Neuroplasticity is highest in childhood, and the visually deprived brain is likely to be most receptive to alternative sensory stimulation in this age group.
2. The BrainPort is non-invasive.
3. Other than gene therapy for Leber's Congenital Amaurosis, there are no alternatives to restoring vision for the blind children at this time.
4. The BrainPort already has CE Mark approval and pending FDA approval (final safety study documents submitted to the FDA August 2013), and should be available for purchase by 2014, at least in Europe and Canada. Whether the device could be useful in a pediatric population is an important clinical question.
5. The relation of the anticipated benefit to the risk presented by the study is at least as favorable to the subjects as that provided by available alternative approaches (blind training).

ELIGIBILITY:
Inclusion Criteria:

Blind Children:

1. Between the age of 4 and 17.
2. Blind (documented visual acuity of light perception or worse) in both eyes from an eye care provider.
3. Able to understand and sign the Informed Consent and Assent form.
4. Able to understand the training and rehabilitation protocols involved in the study.
5. Willing to use the BrainPort device.
6. Able to undergo functional neuroimaging tests

Sighted Children:

1. Between the age of 4 and 17.
2. Sighted in both eyes from an eye care provider.
3. Able to understand and sign the Informed Consent and Assent form.
4. Able to understand the training and rehabilitation protocols involved in the study.
5. Willing to use the BrainPort device.
6. Able to undergo functional neuroimaging tests

Exclusion Criteria:

Blind Children:

1. Current oral health problems as determined by the subject's history, and an examination of the oral cavity performed by a member of the study team. Subject is excluded if any of the following conditions are met:

   1. A history of injury to the tongue resulting in impaired sensation or use of the tongue.
   2. Visible open lesions, cold sores, abrasions, blisters, or rash on the tongue.
   3. Oral surgery or dental work in the past 3 months or anticipated to occur for the duration of participation in the study (does not include routine dental health exams/cleanings).
   4. Piercing on the tongue.
   5. Performance better than 20/5000 on the FrACT acuity test (same visual criteria as FDA safety study).
2. Known neuropathies of tongue or skin tactile system.
3. Unwilling or unable to adhere to all study requirements, including completion of the training period, evaluation tests and follow up visits.
4. Implanted electrical medical devices such as pacemakers.
5. Known allergies to nickel, gold or other components of stainless steel.
6. Patients who are 18 years and older or younger than 4.
7. Women who are pregnant or breast feeding will not be able to participate in this study (as indicated by a positive pregnancy test).
8. Children with neurodevelopmental disorders (e.g., autism, learning disabilities) or congenital brain malformations will be excluded from participation.
9. Cortical blindness from any cause.
10. Claustrophobia that would prevent functional neuroimaging (for those subjects undergoing neuroimaging only).
11. Obesity preventing placement in MRI scanner (for those subjects undergoing neuroimaging only).
12. Presence of any foreign metal in the body with the exception of dental fillings.
13. Implanted metallic or ferromagnetic objects (aneurysm clip, ear implant, IUD, shrapnel or metallic fragments in or on the body or eyes, neuro-stimulators, or other metal devices).

Sighted Children:

1. Current oral health problems as determined by the subject's history, and an examination of the oral cavity performed by a member of the study team. Subject is excluded if any of the following conditions are met:

   1. A history of injury to the tongue resulting in impaired sensation or use of the tongue.
   2. Visible open lesions, cold sores, abrasions, blisters, or rash on the tongue.
   3. Oral surgery or dental work in the past 3 months or anticipated to occur for the duration of participation in the study (does not include routine dental health exams/cleanings).
   4. Piercing on the tongue.
2. Known neuropathies of tongue or skin tactile system.
3. Unwilling or unable to adhere to all study requirements, including completion of the training period, evaluation tests and follow up visits.
4. Implanted electrical medical devices such as pacemakers.
5. Known allergies to nickel, gold or other components of stainless steel.
6. Patients who are 18 years and older or younger than 4.
7. Women who are pregnant or breast feeding will not be able to participate in this study (as indicated by a positive pregnancy test).
8. Children with neurodevelopmental disorders (e.g., autism, learning disabilities) or congenital brain malformations will be excluded from participation.
9. Cortical blindness from any cause.
10. Claustrophobia that would prevent functional neuroimaging (for those subjects undergoing neuroimaging only).
11. Obesity preventing placement in MRI scanner (for those subjects undergoing neuroimaging only).
12. Presence of any foreign metal in the body with the exception of dental fillings.
13. Implanted metallic or ferromagnetic objects (aneurysm clip, ear implant, IUD, shrapnel or metallic fragments in or on the body or eyes, neuro-stimulators, or other metal devices).

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2014-01; Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Mitchell, MD, Principal Investigator — Assistant Professor of Ophthalmology
Locations (1):
- UPMC Eye Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We were unable to enroll sighted children into the study
Period: Overall Study
Arm/Group | Blind Children
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Blind Children
Number analyzed (Participants) | 9
Age, Continuous [Mean (Full Range); unit: years] | 9.67 [5 to 17]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: not collected
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Evaluate BrainPort Device
Description: The efficacy endpoint for this study is a statistical analysis of subjects' improvement over baseline in any of the following areas: light detection, light localization, movement perception (BaGA testing), and standardized object recognition tasks after use of the BrainPort. The mean data reported is the average percentage that participants were able to successfully complete the tested tasks over the 5 visits.
Time Frame: 5 visits over the course of approximately 2 weeks
Measure: Mean (Standard Deviation); unit: percentage of accuracy completing task
Arm/Group | Blind Children
Number analyzed (Participants) | 9
percentage of accuracy completing task
  object identification | 77.36 (20.83)
  object location | 65.47 (27.82)
  light perception | 77.99 (34.99)
  location resolution | 38.0 (20.09)
  BaGA testing | 27.86 (15.14)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Blind Children
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT03002597/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/97/NCT03002597/ICF_001.pdf